CLINICAL TRIAL: NCT02314494
Title: A Feasibility Study of an Interactive, Educational Programme to Facilitate Proactive Assessment of Overweight Risk During Infancy
Brief Title: Proactve Assessment of Overweight Risk During Infancy
Acronym: ProAsk
Status: Completed | Type: Observational
Sponsor: Anglia Ruskin University (Other)
Collaborators: University of Nottingham (Other); University of Lincoln (Other); University of Cambridge (Other); Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: FHSCE001
Record Dates: First submitted 2014-12-05; First posted 2014-12-11 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2015-12

CONDITIONS: Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Infants at risk: Infants identified as at risk of obesity using the ProAsk intervention
  Interventions: Behavioral: ProAsk
- Infants not at risk: Infants identified as not at risk of obesity using the ProAsk intervention.

INTERVENTIONS:
Behavioral: ProAsk — The intervention is a computer programme ProActive Assessment of Overweight Risk to identify infants at risk of developing childhood overweight and obesity. Parents of infants identified as at risk will be offered strategies for prevention by UK health visitors (public health nurses)
  Groups: Infants at risk

SUMMARY:
Children who are above healthy weight are more likely to be ill and to miss time off school. Being overweight in childhood can also sow the seeds for health problems in later life such as heart disease and diabetes. Most overweight children become overweight adults. One solution is to try to prevent children becoming overweight by intervening very early in life. The risk factors for childhood overweight are known and this project aims to facilitate parents' (and other carers') understanding about this for their infant and to enable them to access intervention. UK health visitors (public health nurses) will use an interactive, multimedia programme (Proactive Assessment of Overweight Risk during infancy (ProAsk)), with parents to calculate their infant's risk and to discuss strategies for risk reduction as appropriate. Health visitors will be trained to communicate obesity risk and in Motivational Interviewing techniques to enable them to offer intervention to parents of infants identified as at risk.

A feasibility study of ProAsk will take place in two health provider organisations in the UK. The purpose of this is to a) determine the acceptability and utility of the ProAsk intervention with health visitors and parents and b) gather information to inform the trial design and data collection procedures for a future Randomised Controlled Trial (RCT).

DETAILED DESCRIPTION:
Globally, overweight and obesity is a significant public health issue affecting more than 40 million children under the age of five in 2011. There is broad agreement around the aetiology of childhood overweight and obesity and risk factors have been identified prenatally, during pregnancy and early infancy. Clearly, from the point of view of the infant, risk factors that are present prenatally or during pregnancy are non-modifiable but those identified during infancy are potentially modifiable. Between 25%-33% of infants gain weight more rapidly than desirable during the first 6 months of life and this is the strongest risk factor for childhood overweight at 3 years. Rapid weight gain is potentially modifiable with interventions to facilitate better infant diet, feeding practices and exposure to physical activity. To facilitate identification of infants that might be at greater risk of developing childhood overweight and obesity a number of models have been developed. The Infant Risk of Obesity Checklist (IROC) was developed by the research team using data from the Millennium Cohort Study (MCS) and Avon Longitudinal Study of Parents and Children (ALSPAC) to potentially screen infants at 4 months of age for risk factors for childhood overweight and obesity at 3 years. However, it has not yet been tested in clinical practice.

Concerns have been expressed about using tools developed from the epidemiological literature to identify overweight and obesity risk where there are few effective evidence-based interventions for those affected. There is evidence that complex interventions targeting diet and feeding delivered to parents of infants <2 years old show some positive intervention effects on feeding practices and physical activity, although many of these interventions do not tackle the psycho-emotional aspects of feeding and are not underpinned by behavioural change theory. The impact on weight outcomes is less certain, and in some cases this may be due to intervention components and behaviour change techniques targeted at the parent rather than infant level. Universal eligibility for overweight and obesity prevention is costly and may be unnecessary for those with a low baseline risk. However, targeting of certain groups where overweight and obesity is more prevalent (for example, lower socio-economic status, minority ethnic groups) has raised concerns around stigmatisation. Preliminary work with parents/legal guardians/carers suggests that targeting may be appropriate provided the person conveying the information has appropriate knowledge and sensitivity. his suggests a novel approach to such discussions is needed. Digital technologies are being used to provide information to patients about health care related areas. The findings of a recent review suggest that interactive multimedia programmes have the capacity to facilitate communication between health professionals and patients, but further research in this field is needed.

A pragmatic research design is planned with three linked phases. The first involved the development of an interactive multimedia programme, namely ProActive Assessment of Overweight Risk during Infancy (ProAsk) which includes the IROC and a therapeutic wheel, to facilitate health professionals' discussions with parents/legal guardians/carers about overweight risk and prevention during infancy. This phase is a feasibility study of the ProAsk intervention with parents/legal guardians/carers and health professionals. The study will gather information to inform the trial design and data collection procedures for a Randomised Controlled Trial (RCT) of overweight risk identification and intervention during infancy by UK health visiting teams.

The third phase will be conducted at the end of the feasibility trial .Qualitative work will be undertaken to determine the acceptability and utility of ProAsk with the health professionals working in a health visiting team and parents/legal guardians/carers.

ELIGIBILITY:
Inclusion Criteria:

* Parents/legal guardians/carers of infants aged 6-8 weeks
* First or subsequent born infants

Exclusion Criteria:

* Parents/legal guardians/carers of infants with known medical conditions requiring special diets
* Mothers who have a diagnosis of post-natal depression (PND) or who score moderate PND or above on health visitor applied screening tools (EPDS >13) (PHQ-9 >10) or anxiety (GAD-7 score >10)
* Infants born <32 weeks gestation
* Infants born 32-40 weeks whose birth weight is less than 2nd centile
* Infants born at term (40 weeks) who weigh less than 2.5 kg
* Parents/legal guardians/carers who lack sufficient command of English to complete questionnaires where no face to face translation is available

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants 6-8 weeks old living in the study areas (Cambridshire and Nottingham City)
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2015-05; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Acceptability and utility of the ProAsk intervention | 12 months
  Recruitment, retention, intervention delivery and attrition rates. Proportion of infants calculated as at risk of developing childhood overweight/obesity

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Redsell, PhD, Study Director — Anglia Ruskin University
Locations (2):
- United Kingdom (2):
  - Cambridgeshire Community Services, Cambridgeshire
  - Nottingham City Care Partnership, Nottingham

REFERENCES:
- [Derived] Rose J, Glazebrook C, Wharrad H, Siriwardena AN, Swift JA, Nathan D, Weng SF, Atkinson P, Ablewhite J, McMaster F, Watson V, Redsell SA. Proactive Assessment of Obesity Risk during Infancy (ProAsk): a qualitative study of parents' and professionals' perspectives on an mHealth intervention. BMC Public Health. 2019 Mar 12;19(1):294. doi: 10.1186/s12889-019-6616-5. PMID 30866879
- [Derived] Redsell SA, Rose J, Weng S, Ablewhite J, Swift JA, Siriwardena AN, Nathan D, Wharrad HJ, Atkinson P, Watson V, McMaster F, Lakshman R, Glazebrook C. Digital technology to facilitate Proactive Assessment of Obesity Risk during Infancy (ProAsk): a feasibility study. BMJ Open. 2017 Sep 6;7(9):e017694. doi: 10.1136/bmjopen-2017-017694. PMID 28882926